CLINICAL TRIAL: NCT06618248
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Clinical Trial to Evaluate the Efficacy and Safety of the Sirolimus-coated Spiral Balloon Catheter for the Treatment of Coronary Bifurcation Lesions
Brief Title: Efficacy and Safety of Sirolimus-Coated Spiral Balloon for Coronary Bifurcation Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dongguan TT Medical (Industry)
Collaborators: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCB-CTP-B-V1
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Coronary Bifurcation Lesion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus-coated spiral balloon (SuperFlow®) (Experimental): A PTCA spiral balloon catheter with sirolimus coating (3ug/mm^2) on balloon surface
  Interventions: Combination Product: Sirolimus coated balloon angioplasty
- Paclitaxel-coated balloon (Bingo™） (Active Comparator): A PTCA balloon catheter with paclitaxel coating (3ug/mm^2) on balloon surface
  Interventions: Combination Product: Paclitaxel coated balloon angioplasty

INTERVENTIONS:
Combination Product: Sirolimus coated balloon angioplasty — This study involves the use of a Sirolimus-Coated Balloon (SCB) for the treatment of coronary artery disease, specifically targeting coronary bifurcation lesions. The SCB is coated with sirolimus, an antiproliferative drug that helps to prevent restenosis by inhibiting smooth muscle cell proliferation. The balloon is inflated at the target lesion site, delivering the drug directly to the arterial wall. This intervention aims to achieve vessel dilation while reducing the risk of restenosis, providing a potential alternative to stent placement.
  Arms: Sirolimus-coated spiral balloon (SuperFlow®)
Combination Product: Paclitaxel coated balloon angioplasty — This study involves the use of a Paclitaxel-Coated Balloon (PCB) for the treatment of coronary artery disease, specifically targeting coronary bifurcation lesions. The PCB is coated with paclitaxel, an antiproliferative drug that helps to prevent restenosis by inhibiting smooth muscle cell proliferation. The balloon is inflated at the target lesion site, delivering the drug directly to the arterial wall. This intervention aims to achieve vessel dilation while reducing the risk of restenosis, providing a potential alternative to stent placement.
  Arms: Paclitaxel-coated balloon (Bingo™）

SUMMARY:
This is a multicenter, prospective randomized controlled study to evaluate the safety and effectiveness of Sirolimus-coated spiral balloon (SuperFlow®) versus Paclitaxel-coated balloon (Bingo™) in the treatment of coronary bifurcation lesions.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled, non-inferiority trial conducted across 13-20 sites. The study aims to enroll 280 patients with true coronary bifurcation lesions in native coronary arteries.

Eligible patients will be randomized in a 1:1 ratio to receive either the Sirolimus-coated spiral balloon (SuperFlow®) or the Paclitaxel-coated balloon (Bingo™), following a site-specific blocked randomization schedule.

All participants will be screened based on the trial's predefined inclusion and exclusion criteria. Data and imaging will be collected during the index procedure and at the predefined 9-month clinical follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85 years, regardless of gender.
* Patients must voluntarily participate in the study and sign an informed consent form.
* Patients must demonstrate sufficient adherence to the study protocol and agree to follow-up visits at 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days) post-procedure, with angiography required at 9 months (±30 days).
* Patients must have evidence of myocardial ischemia.
* Angiographically confirmed primary coronary bifurcation lesions (Medina classification non-0, 0, 1) with branch stenosis ≥70% (estimated visually).
* Patients suitable for PCI where the branch lesion is not expected to require stenting; stenting is planned for the main vessel, with DCB used on the branch. It is recommended to treat the branch with DCB first, followed by main vessel stenting.
* Residual stenosis ≤50% after pre-treatment of the branch lesion, TIMI 3 flow, with no dissection or only A or B grade dissection. C grade dissections should be carefully considered by the investigator before deciding, and are generally not included.
* The diameter of the branch vessel must be between 2.0 mm and 4.0 mm, with a lesion length ≤40 mm.

Exclusion Criteria:

* Patients with bleeding disorders or active gastrointestinal ulcers, those who have had a stroke within the past 6 months, or those who are expected to be intolerant to dual antiplatelet therapy post-intervention.
* Patients with severe renal insufficiency (creatinine level > 3.0 mg/dL or 265.2 µmol/L) and/or end-stage renal disease requiring dialysis.
* Patients in cardiogenic shock.
* Patients who have experienced a myocardial infarction within the week prior to enrollment.
* Patients with severe congestive heart failure or NYHA class IV severe heart failure.
* Patients with severe valvular heart disease.
* Patients who have undergone heart transplantation.
* Patients with a life expectancy of less than 1 year.
* Patients currently participating in other drug or device clinical trials that have not yet reached the primary endpoint.
* Patients with contraindications to taking aspirin and/or clopidogrel and/or ticagrelor.
* Patients known to be allergic to paclitaxel, rapamycin, contrast agents, etc.
* Pregnant or breastfeeding women, those with plans to conceive within the year, or those unwilling to use effective contraception.
* Target vessels that are completely occluded, severely calcified, have >45° angulation, or are non-protected left main lesions.
* Non-target lesions that cannot be treated prior to or fail to be treated successfully before addressing the target lesion.
* Target lesions in branch vessels that are in-stent restenosis.
* Other patients deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Diameter stenosis (%) | 6 months (±30 days)
  Percentage of target vessel stenosis per angiographic measurement at 6 months follow up

SECONDARY OUTCOMES:
Interventional success rate | Immediate post procedure (device and lesion success), and up to 7 days post-procedure (clinical success)
  Including device success, lesion success, and clinical success
  Device Success: Includes successful delivery of the device and successful treatment.
  Successful Delivery: Successful delivery of the designated device to the lesion and release, with the delivery system retracting smoothly. Successful Treatment: Immediately post-procedure, residual stenosis of the target lesion is less than 50% with TIMI grade 3 flow (visual assessment).
  Lesion Success: After any interventional treatment, residual stenosis of the target lesion is less than 50% with TIMI grade 3 flow (visual assessment).
  Clinical Success: Based on lesion success, no major adverse cardiac events occurred during hospitalization (up to 7 days post-procedure).
Quantitative Flow Ratio (QFR) | 9 months (±30 days)
  In the presence of stenotic lesions in the coronary artery, the ratio of the maximum blood flow that the artery can deliver to the myocardial region to the maximum blood flow that could theoretically be obtained in that region under normal conditions.
Rate of restenosis | 9 months (±30 days)
  Coronary angiography results showing a diameter stenosis of ≥50% are considered indicative of restenosis.
Late lumen loss (LLL) | 9 months (±30 days)
  The difference between the minimum lumen diameter of the target lesion segment immediately post-procedure and the minimum lumen diameter of the same segment during the angiographic follow-up at 9 months post-procedure.
Target lesion revascularization (TLR) | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days)
  Including repeat PCI with stent implantation, balloon angioplasty, plaque atherectomy, or coronary artery bypass grafting (CABG)
Target vessel revascularization (TVR) | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days)
  Including repeat PCI with stent implantation, balloon angioplasty, plaque atherectomy, or CABG
Target lesion failure (TLF) rate | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days)
  Including cardiac death, target vessel-related myocardial infarction, and target lesion revascularization
Thrombotic event rate | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days)
  Rate of thrombosis
Major adverse cardiac events (MACE) rate | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days)
  Including all-cause death, all myocardial infarctions, and all repeat revascularizations
Adverse events (AEs) and serious adverse events (SAEs) rate | 1 month (±7 days), 6 months (±14 days), 9 months (±30 days), 12 months (±30 days), and 24 months (±30 days)
  Rate of AEs or SAEs
Device defect rate | Immediate post procedure
  Rate of device defect

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wu, MD, PhD, Study Chair — Dongguan TT Medical
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No